CLINICAL TRIAL: NCT02797431
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Study of IL-7 to Restore Absolute Lymphocyte Counts in Sepsis Patients
Brief Title: Immune Reconstitution of Immunosuppressed Sepsis Patients
Acronym: IRIS-7a
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: failure of supply of test product
Sponsor: University Hospital, Limoges (Other)
Collaborators: Revimmune (Industry); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I14037 IRIS-7a
Record Dates: First submitted 2016-02-24; First posted 2016-06-13 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Severe Sepsis With Septic Shock
MeSH Terms: interventions — Interleukin-7; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CYT107 high frequency (Experimental): Patients will receive Interleukin-7 (CYT107 liquid solution) at 10µg/kg twice a week for 4 weeks
  Interventions: Drug: Interleukin-7
- CYT107 low frequency (Experimental): Patients will receive Interleukin-7 (CYT107 liquid solution) at 10µg/kg twice a week for the first week, followed by CYT107 and Placebo once a week for the three following weeks
  Interventions: Drug: Interleukin-7; Drug: Placebo
- Control (Placebo Comparator): Patients will receive Placebo (NaCl 0.9%) twice a week for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interleukin-7 — IM administration of CYT107 recombinant glycosylated human IL-7 (SC administration for patients with INR>2.5 or platelet count < 35,000
  Other Names: CYT 107
  Arms: CYT107 high frequency; CYT107 low frequency
Drug: Placebo — IM administration of Placebo (SC administration for patients with INR>2.5 or platelet count < 35,000
  Other Names: NaCl 0.9%
  Arms: CYT107 low frequency; Control

SUMMARY:
A multicenter, randomized, double-blinded, placebo-controlled study of two dosing frequencies of recombinant Interleukin-7 (CYT107) treatment to restore absolute lymphocyte counts in sepsis patients; IRIS-7A (Immune Reconstitution of Immunosuppressed Sepsis patients).

A parallel study will be performed in United State of America to allow a common statistical analysis of the primary end points and analysis for the enrolled patient population.

DETAILED DESCRIPTION:
Sepsis is the leading cause of death in critically ill patients in most intensive care units in Europe and the US. Recently, evidence has accumulated that sepsis progresses from a state of hyper-inflammation to a state of immunosuppression. This immunosuppressive phase is characterized by increased incidence of secondary infections often with relatively avirulent opportunistic type pathogens. Currently, new therapeutic approaches to sepsis are occurring using immuno-adjuvants that boost host immunity. One of the most promising agents Interleukin-7 is an essential, non-redundant, pluripotent cytokine produced mainly by bone marrow and thymic stromal cells that is required for T-cell survival.In addition to its anti-apoptotic properties, IL-7 induces potent proliferation of naïve and memory T-cells potentially supporting replenishment of the peripheral T-cell pool which is severely depleted during sepsis. These effects were confirmed in clinical trials at the National Cancer Institute and in HIV+ patients.

This clinical study will test the ability of IL-7 to restore the absolute lymphocyte counts in septic patients who have markedly reduced levels of circulating lymphocytes. An effect already confirmed in preclinical models of sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of age ≥ 18 yrs and older but < 80 yrs
2. Patients with persistent suspected sepsis at 48-120 hrs after admission
3. Two or more criteria for the systemic inflammatory response syndrome (SIRS) (see reference #19 for SIRS criteria) and a clinically or microbiologically suspected infection.
4. At least one organ failure as defined by a SOFA score of ≥2 at any time point during the 48-120 hrs after admission to the ICU
5. Requirement of vasopressor treatment as follows: i) epinephrine or norepinephrine at ≥ 0.05 µg/kg/min ideal body weight; ii) vasopressin, or iii) dopamine at ≥ 4-5 μg/kg/min ideal body weight, continuously for 4 hrs or more, provided that at least 20 ml/kg of ideal body weight of crystalloid or an equivalent volume of colloid was administered during the 24-hour interval surrounding the start of vasopressor treatment, to maintain systolic pressure ≥ 90 mmHg or a mean arterial pressure ≥ 60 mmHg at any time point during their sepsis course preceding enrollment into the IL-7 study.
6. Lymphopenia with an absolute lymphocyte count ≤ 900 cells/mm3 at either the day of consent or the day prior to consent during their ICU stay.
7. Predicted length of stay in the ICU of up to two weeks after starting drug therapy treatment in the trial
8. Ability to obtain a signed informed consent from patient or LAR consent.

Exclusion Criteria:

1. Cancer with current chemotherapy or radiotherapy and/or .receipt of chemotherapy or radiotherapy within the last 6 weeks
2. Cardiopulmonary resuscitation within the previous 4 weeks without objective evidence of full neurologic recovery) or patients who have minimal chance of survival and are not expected to live > 3-5 days as defined by an APACHE II score of ≥ 35 at time of consideration for study eligibility
3. Patients with a history of or who currently have evidence of autoimmune disease including for example: myasthenia gravis, Guillain Barre syndrome, systemic lupus erythematosis, multiple sclerosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's etc.
4. Patients who have received solid organ transplant or bone marrow transplant
5. Patients with active or a history of acute or chronic lymphocytic leukemia
6. AIDS-defining illness (category C) diagnosed within the last 12 months prior to study entry
7. History of splenectomy
8. Any hematologic disease associated with hypersplenism, such as thalassemia, hereditary spherocytosis, Gaucher's Disease, and autoimmune hemolytic anemia
9. Pregnant or lactating women
10. Participation in another investigational interventional study within the last 6 months prior to study entry, with the exception of studies aimed at testing sedation products belonging to standard of care such as Propofol, Dexmedetomidine, Midazolam.
11. Patients receiving immunosuppressive drugs, e.g., TNF-alpha inhibitors, for rheumatoid arthritis, inflammatory bowel disease or any other reason, or systemic corticosteroids other than hydrocortisone at a dose of 300 mg/day
12. Patients receiving concurrent immunotherapy or biologic agents including: growth factors, cytokines and interleukins, (other than the study medication); for example IL-2,growth factors, interferons, HIV vaccines, immunosuppressive drugs, hydroxyurea, immunoglobulins, adoptive cell therapy
13. Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
White blood count | day 1 to Day 42
  Number of patients with absolute lymphocyte counts (Multiply the Lymphocytes percentage above by the total number White Blood Count) increased by more than 50% from baseline at Day 42 Kinetic of immune restoration through weekly measures of Absolute Lymphocyte Counts
lymphocyte percentage | Day 1 to Day 42
  Number of patients with absolute lymphocyte counts (Multiply the Lymphocytes percentage above by the total number White Blood Count) increased by more than 50% from baseline at Day 42 Kinetic of immune restoration through weekly measures of Absolute Lymphocyte Counts
Incidence of treatment-Emergent Adverse Events | Day 1 to Day 42
  Clinical occurrence of adverse events (AEs) and serious adverse events (SAEs) during the duration of the study period ending day 42, as assessed by DAIDS (2.0)
Mortality | Day 60
Mortality | Day 190
Mortality | Day 180
Mortality | Day 360

SECONDARY OUTCOMES:
CYT107 Pharmacokinetic Cmax | Day 1 and Day 22
  CYT107 PK: Measure of Peak plasma concentration "Cmax" at Day 1 and Day 22
CYT107 Pharmacokinetic AUC | Day 1 and Day 22
  CYT107 PK: Measure of Area under plasma concentration versus time curve at day 1 and day 22
CYT107 Pharmacokinetic half life | Day 1 and Day 22
  CYT107 PK: Measure plasma concentration half life at day 1 and day 22
Quantification of positive binding antibodies against CYT107 | Day 1, Day 11, Day 22, Day 60, Day 180 and Day 360
  number of patients with positive binding antibodies against CYT107 at Day 1, Day 11, Day 22, Day 60, Day 180 if Day 60 is positive and Day 360 if Day 180 is positive.
Specific CYT107 neutralizing antibodies | Day 1, Day 11, Day 22, Day 60, Day 180 and Day 360
  Number of patients with CYT107 neutralizing antibodies if positive binding antibodies against CYT107 is detected.
Incidence of hospital acquired secondary infections | Day 42
  Incidence of hospital acquired secondary infections at Day 42
SOFA score | Day 0 Day 4, Day 8, Day 15, Day 22, Day 29
  SOFA score at Day 0 Day 4, Day 8, Day 15, Day 22, Day 29.
APACHE II score | Day 0, Day 4, Day 8, Day 15, Day 22, Day 29
  APACHE II score at Day 0, Day 4, Day 8, Day 15, Day 22, Day 29.
CYT107 Pharmacodynamic | Day 1, Day 8, Day 15, Day 22, Day 29
  CYT107 effects on cell counts:
  T-CD4+, T-CD8+, T-CD127+ (IL-7R), monocyte HLA-DR+

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FRANCOIS, DM, Principal Investigator — University Hospital, Limoges
Locations (3):
- France (3):
  - CHU LIMOGES Service de Réanimation, Limoges
  - Hospice Civil de Lyon - Hôpital Edouard Herriot - Service de Réanimation Médicale, Lyon
  - Hopital Lariboisière - Service d'anesthésie-réanimation, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Francois B, Jeannet R, Daix T, Walton AH, Shotwell MS, Unsinger J, Monneret G, Rimmele T, Blood T, Morre M, Gregoire A, Mayo GA, Blood J, Durum SK, Sherwood ER, Hotchkiss RS. Interleukin-7 restores lymphocytes in septic shock: the IRIS-7 randomized clinical trial. JCI Insight. 2018 Mar 8;3(5):e98960. doi: 10.1172/jci.insight.98960. PMID 29515037